CLINICAL TRIAL: NCT05682274
Title: The Effect of Placement of the Apical Margin of the Restoration in the Treatment of Gingival Recession Associated With Non-carious Cervical Lesion With Combined Restorative and Periodontal Therapy
Brief Title: Effect of Restoration Margin Level in the Treatment of Gingival Recession Associated With Non-carious Cervical Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-21071282-050.99-108427
Record Dates: First submitted 2022-12-25; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Gingival Recession, Localized
Keywords: Gingival recession; Tooth abrasion; Composite resin; Connective tissue graft; Dental sensitivity
MeSH Terms: conditions — Gingival Recession; Tooth Abrasion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Partial restoration with the apical border at the level of CEJ in combination with CAF+CTG
  Interventions: Procedure: Partial restoration approach combined with CAF+CTG
- Group II (Active Comparator): Partial restoration with the apical border within 1 mm apical to the CEJ.
  Interventions: Procedure: Partial restoration approach combined with CAF+CTG

INTERVENTIONS:
Procedure: Partial restoration approach combined with CAF+CTG — The location of the CEJ prior to the restorative treatment was identified using the method developed by Zuchelli et al. 2006. The placement of the apical margin of the restoration was performed either at the level of estimated cementoenamel junction (CEJ) or within 1 mm apical to the CEJ. Two weeks after the restorative treatment, all recession defects were treated with CAF combined with CTG.

SUMMARY:
The aim of this randomized, parallel-group clinical trial was to compare the 1-year periodontal, root coverage, esthetic, and patient-centered outcomes of the partial restoration placement with different apical margin levels combined with coronally advanced flap (CAF) plus connective tissue graft (CTG) in the treatment of isolated gingival recessions associated with non-carious cervical lesions (NCCL). Forty patients with single gingival recessions (RT1 gingival recessions and class B+ NCCL) were randomly allocated to either placement of restoration apical margin at the level of estimated cementoenamel junction (CEJ) or within 1 mm apical to the CEJ. Two weeks after the restorative treatment, all recession defects were treated with CAF combined with CTG. Periodontal measurements were taken at baseline, and 3, 6, and 12 months postoperatively. Patient-centered outcomes were evaluated at baseline, and 7, and 15 days, 6, and 12 months postoperative follow-ups. Modified root closure aesthetic score (mRES) was used to assess aesthetics at 6 and 12 months follow-ups.

DETAILED DESCRIPTION:
Gingival recessions associated with non-carious cervical lesions (NCCL) involving the CEJ area, which form a combined defect (CD), can lead to complex soft tissue management during periodontal plastic surgeries and result in poor clinical/aesthetic outcomes. Since CD encompasses both hard and soft tissue loss, different periodontal/restorative multidisciplinary protocols have been suggested to treat this challenging situation. Reconstruction of the coronal portion of NCCL with a resin composite filling (partial restoration approach) before the surgical procedure has been suggested to present favorable and predictable outcomes in the treatment of gingival recessions associated with NCCL. For the partial restoration approach, two different protocols to restore the most coronal zone of the NCCL have been proposed according to the extension of the apical margin of the restoration, which are the placements at the level of CEJ or within 1 mm apical to the CEJ. Both approaches have some advantages and disadvantages. After root coverage procedures, if complete closure has been achieved, placing the apical restoration margin at the estimated CEJ level would allow the gingival margin to contact only the root surface and not cover the apical part of the restoration. However, in cases with incomplete root coverage, the placement of the restoration border 1 mm apically of the CEJ could prevent the formation of a gap between the gingival margin and the apical border of the restoration that results in esthetic compromises, and the persistence of dentin hypersensitivity. However, there is no study in the literature comparing these two different locations of the apical border of the restoration in periodontal/restorative combined therapy. Therefore, the aim of this study was to compare the 1-year periodontal, root coverage, esthetic, and patient-centered outcomes of the partial restoration placement with different apical margin levels combined with CAF plus CTG in the treatment of isolated gingival recessions associated with NCCL.

Material and Methods

This randomized, parallel-group clinical study recruited 40 systemically healthy patients, who were admitted to Gazi University Faculty of Dentistry, Department of Periodontology with complaints of sensitivity and aesthetic problems due to gingival recession. The patients were randomly assigned to the study groups: group I, partial restoration with the apical border at the level of CEJ in combination with CAF+CTG; group II, partial restoration with apical border within 1 mm apical to the CEJ.

The location of the CEJ prior to the restorative treatment was identified using the method developed by Zuchelli et al. 2006.

The gingival margin to the most coronal of the NCCL, as well as the width and depth of the NCCL, were measured before and after the restorative treatment. Periodontal parameters were measured with a periodontal probe (UNC 15) at baseline, and 3, 6, and 12 months postoperatively. Plaque index (PI), gingival index (GI), probing depth (PD), bleeding on probing (BOP), clinical attachment level (CAL), recession depth (RD), recession width (RW), keratinized tissue width (KTW), and gingival thickness (GT) were all measured and recorded.

The flap thickness, graft width, height, and thickness were measured during the procedures. On the 7th and 14th days, postoperative pain, sensitivity, and aesthetic scores were determined using a 0-10 visual analog scale in the patient-based evaluation (VAS). Furthermore, the modified root closure aesthetic score (mRES) was used to assess aesthetics objectively at the 6 and 12-month follow-ups.

Restorative procedure

The defect surface was roughened with 37% orthophosphoric acid before being washed and dried while still moist. The adhesive resin was then applied to the surface as directed by the manufacturer. 3M ESPE, Deutchland GmbH, Neuss, GERMANY (Single Bond Universal). Finally, a 2 mm thick restorative material (Tetric Evo Ceram, Ivoclar Vivadent, Schaan, Liechtenstein) was applied to the restoration area and polymerized by applying light for 20 seconds. Finally, the restoration surfaces were polished, and the restoration margins were checked with a blunt-tipped probe. Two weeks later, the patients underwent periodontal surgery.

Surgical Technique

Following the CEJ, a sulcular incision was made in the gingival margin of the tooth using a microblade, and a horizontal incision was made from the tooth with recession to the adjacent teeth. The vertical incision towards the apex and the horizontal incision was then intersected. The muscle attachments were cut after gentle elevation. A split-full-split thickness flap was raised up beyond the MGJ. A gentle root debridement was performed using a sharp curette up to 1 mm from the bone crest. CPF technique designed by Zuchelli and De Sanctis (2000) was performed. Then the flap was elevated and CTG, which was fixed with the coronal border at the level of restored CEJ, was sutured. The flap was stabilized and sutured 1-2 mm above the restored CEJ with a 6/0 Teflon suture.

Obtaining CTG from Palatinal Mucosa

The graft margins were determined with a 15C scalpel by making two horizontal incisions parallel to the palatal midline of the preferred donor area and two vertical incisions perpendicular to them, 2 mm away from the apical of the gingival margin of the teeth so that the distal extension of the incision ends at the mesial border of the first molar. The graft's epithelial surface was removed extra orally (0.3-0.5 mm) with the reflection of the scalpel tip visible. The graft was de-epithelialized and placed in a petri dish with physiological saline.

Care was taken to ensure that the was de-epithelialized approximately 1 mm thick, similar to conventional free gingival grafts. By controlling the bleeding in the donor area, a hemostatic sponge was sutured using the vertical cross-suture technique.

Post-operative Care

The patients were recommended not to brush the operation area for 2 weeks and were instructed to use 0.12% CHX (Kloroben, Drogsan Istanbul, Turkey) mouthwash twice a day. For post-operative pain, patients were advised to take 400 mg of the non-steroidal anti-inflammatory drug (ibuprofen) twice a day for 14 days. Sutures were removed 14 days after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Gingival recession of at least 1 mm depth.
* There is no loss of interdental support (RT-1)
* Cervical step greater than 0.5 mm
* Inability to detect CEJ (Class B+)
* Maximum root closure level at the NCCL's deepest point (Type 3)
* Individuals who do not have any systemic disease that would preclude surgery
* Who are not pregnant
* Who are not smokers or who smoke less than 5 cigarettes per day
* Who have a whole mouth plaque and bleeding score of 10%
* Patients who do not require endodontic treatment in the surgical area and do not have tooth mobility;
* Patients who do not require orthodontic treatment;
* Patients who do not have periodontal disease; and
* Patients who do not have restoration and/or filling in the recession area.

Exclusion Criteria:

* Smokers
* Pregnant
* Having a systemic disease that may deteriorate wound healing
* Poor oral hygiene
* Patients with active periodontal disease
* Tooth devitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in gingival recession height | 12 months after the surgery
  Immediately after reconstruction of CEJ, gingival recession height was measured and accepted as baseline value. This value was obtained by the difference between 12th month gingival recession height and baseline recession height

SECONDARY OUTCOMES:
Mean root coverage | 12 months after the surgery
Complete root coverage | 12 months after the surgery
Modified root closure aesthetic score | 12 months after the surgery
  Modified root closure aesthetic score was evaluated six variables. Gingival margin: 0 or 3 points; marginal tissue contour: 0 or 1 point; soft tissue texture: 0 or 1 point; mucogingival junction alignment: 0 or 1 point; gingival colour: 0 or 1 point; restoration/cervical lesion colour: 0 points = colour of restoration or uncovered cervical lesion does not match tooth colour; 3 points = good colour integration. The total higher score means more favorable outcomes.
Dental sensitivity by visual analogue scale | 12 months after the surgery
  This scale is a 10-centimeter horizontal line with scores of 0 and 10 at their ends, where 0 = no sensitivity and 10 = severe sensitivity.
Self-perceived aesthetic satisfaction by visual analogue scale | 12 months after the surgery
  This scale is a 10-centimeter horizontal line with scores of 0 and 10 at their ends, where 0 = no satisfaction and 10 = fully satisfied
Clinical attachment level | 12 months after the surgery
Probing depth | 12 months after the surgery
Soft tissue thickness phenotype | 12 months after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zucchelli G, Gori G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, De Sanctis M. Non-carious cervical lesions associated with gingival recessions: a decision-making process. J Periodontol. 2011 Dec;82(12):1713-24. doi: 10.1902/jop.2011.110080. Epub 2011 May 4. PMID 21542735
- [Result] Yang S, Lee H, Jin SH. A combined approach to non-carious cervical lesions associated with gingival recession. Restor Dent Endod. 2016 Aug;41(3):218-24. doi: 10.5395/rde.2016.41.3.218. Epub 2016 May 2. PMID 27508164
- [Result] Cairo F, Cortellini P, Nieri M, Pilloni A, Barbato L, Pagavino G, Tonetti M. Coronally advanced flap and composite restoration of the enamel with or without connective tissue graft for the treatment of single maxillary gingival recession with non-carious cervical lesion. A randomized controlled clinical trial. J Clin Periodontol. 2020 Mar;47(3):362-371. doi: 10.1111/jcpe.13229. Epub 2020 Jan 7. PMID 31811742
- [Result] de Sanctis M, Di Domenico GL, Bandel A, Pedercini C, Guglielmi D. The Influence of Cementoenamel Restorations in the Treatment of Multiple Gingival Recession Defects Associated with Noncarious Cervical Lesions: A Prospective Study. Int J Periodontics Restorative Dent. 2020 May/Jun;40(3):333-342. doi: 10.11607/prd.4639. PMID 32233184
- [Result] Pini-Prato G, Franceschi D, Cairo F, Nieri M, Rotundo R. Classification of dental surface defects in areas of gingival recession. J Periodontol. 2010 Jun;81(6):885-90. doi: 10.1902/jop.2010.090631. PMID 20450362
- [Result] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093
- [Result] Cairo F, Pini-Prato GP. A technique to identify and reconstruct the cementoenamel junction level using combined periodontal and restorative treatment of gingival recession. A prospective clinical study. Int J Periodontics Restorative Dent. 2010 Dec;30(6):573-81. PMID 20967303
- [Result] Zucchelli G, Testori T, De Sanctis M. Clinical and anatomical factors limiting treatment outcomes of gingival recession: a new method to predetermine the line of root coverage. J Periodontol. 2006 Apr;77(4):714-21. doi: 10.1902/jop.2006.050038. PMID 16584355
- [Result] Santamaria MP, Queiroz LA, Mathias IF, Neves FL, Silveira CA, Bresciani E, Jardini MA, Sallum EA. Resin composite plus connective tissue graft to treat single maxillary gingival recession associated with non-carious cervical lesion: randomized clinical trial. J Clin Periodontol. 2016 May;43(5):461-8. doi: 10.1111/jcpe.12524. Epub 2016 Apr 13. PMID 26847486